CLINICAL TRIAL: NCT01668641
Title: Randomized, Double-blind, Placebo-controlled, Multicenter, Phase II Study to Compare Four Dose Regimens of GLPG0634 Versus Placebo, in Combination With Methotrexate, Administered for 4 Weeks in the Treatment of Subjects With Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate Alone
Brief Title: Dose-ranging Study With GLPG0634 in Methotrexate-refractory Active Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-202
Record Dates: First submitted 2012-08-14; First posted 2012-08-20 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate insufficient responders
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- capsule, 30mg GLPG0634 once a day (Experimental): 3 capsules of 10 mg once a day
  Interventions: Drug: GLPG0634
- capsules, 75mg GLPG0634 once a day (Experimental): 3 capsules of 25mg once a day
  Interventions: Drug: GLPG0634
- capsules, 150mg GLPG0634 once a day (Experimental): 3 capsules of 50mg once a day
  Interventions: Drug: GLPG0634
- capsules, 300mg GLPG0634 once a day (Experimental): 3 capsules of 100mg once a day
  Interventions: Drug: GLPG0634
- capsules, placebo once a day (Placebo Comparator): 3 capsules placebo once a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG0634
  Arms: capsule, 30mg GLPG0634 once a day; capsules, 150mg GLPG0634 once a day; capsules, 300mg GLPG0634 once a day; capsules, 75mg GLPG0634 once a day
Drug: Placebo
  Arms: capsules, placebo once a day

SUMMARY:
* Ninety patients suffering from active rheumatoid arthritis despite continued treatment with methotrexate will be evaluated for improvement of disease activity when taking GLPG0634 (4 different doses will be evaluated) or matching placebo for 4 weeks.
* During the course of the study, patients will also be examined for any side effects that may occur, and the amount of GLPG0634 present in the blood as well as the effects of GLPG0634 on disease- and mechanism of action-related parameters in the blood will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Have active RA as shown by five or more swollen joints (from the 66-joint count), five or more tender joints (from 68-joint count), and a serum CRP ≥1.0 mg/dL;
* Have received methotrexate for 12 weeks or longer and at a stable dose of 7.5 to 25 mg/week for at least 4 weeks prior to screening and willing to continue on this regimen for the duration of the study;
* If taking oral steroids, these should be at a dose ≤10 mg/day of prednisone or prednisone equivalent and stable for at least 4 weeks prior to screening;
* If taking non-steroidal anti-inflammatory drugs (NSAIDs), these must be at a stable dose for at least 2 weeks prior to screening;
* Female subjects must have a negative pregnancy test unless they are surgically sterile or have been post-menopausal for at least one year;
* Women of childbearing potential must use a medically acceptable means of birth control and agree to continue its use during the study and for at least 12 weeks after the last dose of study drug.
* Sexually active men must agree to use a medically acceptable form of contraception during the study and continue its use for at least 3 months after the last dose of study drug; and
* Able and willing to sign the informed consent prior to screening evaluations and agree to schedule of assessments.

Exclusion Criteria:

* Treatment with disease-modifying antirheumatic drugs (DMARDs), other than background methotrexate;
* Current or previous RA treatment with a biological agent, with the exception of biologics administered in a clinical study setting more than six months prior to screening (12 months for rituximab or other B cell depleting agents);
* Previous treatment at any time with a cytotoxic agent, other than methotrexate, before screening;
* Previous use of the study drug GLPG0634;
* Receipt of an intra-articular or parenteral corticosteroid injection within 4 weeks prior to screening;
* Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug as determined by the Investigator;
* Positive serology for HIV1 or 2 or hepatitis B or C, or any history of hepatitis from any cause with the exception of hepatitis A;
* History of any inflammatory rheumatological disorders other than RA;
* History of tuberculosis (TB) infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The number of patients with an ACR20 score at Week 4 as a measure of efficacy | Week 4 (end of treatment visit)
  To preliminary evaluate the efficacy of GLPG0634 compared to placebo in terms of the proportion of subjects achieving an ACR20 response at Week 4

SECONDARY OUTCOMES:
The number of patients with ACR20/50/70 response, time to response and DAS28 score at every visit as a measure of efficacy | From Day -1 up to end of treatment visit (week 4)
  To evaluate the efficacy of GLPG0634 compared to placebo in terms of ACR response criteria at every visit (ACR20, ACR50, ACR70), time to response, and disease status (DAS28[C-reactive protein, CRP]
The number of patients with adverse events, abnormal lab tests, vital signs and ECG as a measure of safety and tolerability | From screening up to 10 days after last dose
  To evaluate the safety and tolerability of GLPG0634 in comparison with placebo in terms of adverse events (AEs), laboratory test abnormalities, vital signs and electrocardiogram (ECG)
The plasma levels of GLPG0634 as a measure of PK | Week 1, week 2 and week 4 visits
  To characterize the pharmacokinetics (PK) of GLPG0634 by measuring the amount of GLPG0634 in the plasma
The plasma levels of GLPG0634 and MTX as a measure of PK | Day -1 and Week 2 or 4 visit (8 hour-sampling)
  To explore the potential interaction of GLPG0634 on MTX by assessing steady state PK in an 8-hour sampling at Day -1 and at Week 2 or Week 4 visit in a subset of patients
The levels of immune- and inflammation-related parameters in plasma as a measure of PD | Day -1, Week 1, week 2 and week 4 visits
  To characterize the pharmacodynamics (PD) of GLPG0634 by measuring the levels of immune- and inflammation-related parameters in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (19):
- Hungary (4):
  - Budai Irgalamsrendi Korhaz, II. Reumatologia Osztaly, Budapest
  - Orszagos Reumatologiai es Fizioterapias Intezet, I. Reumatologia Osztaly, Budapest
  - Markhot Ferenc Korhaz, Reumatologiai Osztaly, Eger
  - Pest Megyei Flor Ferenc Korhaz, Reumatologiai es Fizioterapias Osztaly, Kistarcsa
- IMSP Institutel de Cardiologie, Chisinau, Moldova
- Russia (5):
  - State Healthcare Institution of city Moscow 'City Clinical Hospital #7', Moscow
  - State Healthcare Institution 'Ryazan Regional Cardiology Dispensary', Ryazan
  - Saint-Petersburg State Healthcare Institution 'City Hospital #26', Saint Petersburg
  - Saint-Petersburg State Healthcare Institution 'City Mariinskiy Hospital', Saint Petersburg
  - Municipal Clinical Healthcare Institution 'Medical-Sanitary Unit of Novoyaroslavskiy Oil Refinery', Yaroslavl
- Ukraine (9):
  - Chernivtsi Regional Clinical Hospital, Chernivtsi
  - State Institution 'Institute of Urgent and Recovery Surgery n.a. V.K. Gusaka' of AMS of Ukraine, Donetsk
  - Communal Institution of Healthcare, Kharkiv
  - Institution of Therapy of AMS of Ukraine, Kharkiv
  - State Institution 'Institute of Microbiology and Immunology of AMS of Ukraine', Kharkiv
  - State Institution 'Republican Clinical Hospital of MoH of Ukraine', Kiev
  - Lutsk City Clinical Hospital, Lutsk
  - Vinnytsa Regional Clinical Hospital, Vinnytsa
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhzhia

REFERENCES:
- [Derived] Vanhoutte F, Mazur M, Voloshyn O, Stanislavchuk M, Van der Aa A, Namour F, Galien R, Meuleners L, van 't Klooster G. Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Filgotinib, a Selective JAK-1 Inhibitor, After Short-Term Treatment of Rheumatoid Arthritis: Results of Two Randomized Phase IIa Trials. Arthritis Rheumatol. 2017 Oct;69(10):1949-1959. doi: 10.1002/art.40186. Epub 2017 Aug 31. PMID 28622463